CLINICAL TRIAL: NCT03544099
Title: Pembrolizumab for Nasopharyngeal Carcinoma Patients With Detectable Plasma Epstein-Barr Virus DNA But Without Clinically Detectable Residual Diseases and/or Metastases After Curative Chemoradiation - A Single Arm Phase II Trial
Brief Title: Pembrolizumab for Nasopharyngeal Carcinoma Patients With Detectable Plasma Epstein-Barr Virus DNA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficult to recruit Nasopharyngeal Carcinoma Patients With Detectable Plasma Epstein-Barr Virus DNA
Sponsor: National Health Research Institutes, Taiwan (Other)
Collaborators: National Taiwan University Hospital (Other); Koo Foundation Sun Yat-Sen Cancer Center (Other); Chang Gung Memorial Hospital (Other); Taichung Veterans General Hospital (Other); China Medical University Hospital (Other); Changhua Christian Hospital (Other); National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T1317
Record Dates: First submitted 2018-05-21; First posted 2018-06-01 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: nasopharyngeal carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: Interventional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab for NPC patients (Experimental): Pembrolizumab 200 mg Q3W IV infusion, Day 1 of each 3 week cycle, for 35 cycles
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab 200mg Intravenous Solution
  Other Names: KEYTRUDA

SUMMARY:
This is a single-arm, multi-center, open-label, phase II trial to examine the efficacy of pembrolizumab for prolonging the one-year disease free survival in nasopharyngeal carcinoma patients with solely detectable EBV DNA after curative chemoradiation. Sixty-three patients will be enrolled in the trial.

DETAILED DESCRIPTION:
This phase II study is aimed to prove the efficacy of adjuvant therapy with pembrolizumab for nasopharyngeal carcinoma patients with detectable plasma EBV DNA after curative chemoradiation.

Nasopharyngeal cancer was a malignancy related to Epstein-Barr virus infection. It was a malignancy endemic in Southeast Asia, Taiwan, and China. The primary treatment was chemoradiation. The three-year disease free survival was around 50-60% for locally-advanced (stage IVA, IVB) NPC. Adjuvant chemotherapy after curative chemoradiation is a strategy to improve disease control rate for advanced NPC. However, two phase III trials in Taiwan (TCOG 1394) and China failed to prove its efficacy on improving disease control and overall survival. How to identify patients who are truly at risk is an important question for the therapy of advanced NPC.

Plasma EBV DNA copy number is a biomarker predicting the recurrent risk of nasopharyngeal cancer. A higher level of plasma EBV DNA before chemoradiation is related to a poorer prognosis. A detectable EBV DNA after chemoradiation, which is a hint for occult residual or metastatic disease, is a strong predictor for early recurrence. The relapse free survival at two years for patients with detectable plasma EBV DNA (> 0 copies/mL) was around 20%. The results of other similar trials are summarized on table 1.

Cancer cells escaped from the immune surveillance by several mechanisms. One of them is activating immune inhibitory pathway by "immune checkpoints" . Programmed Death 1 (PD-1) and Programmed Death Ligand 1 (PD-L1) is one immune checkpoint axis to regulate immune response against cancer. Pembrolizumab (MK-3475), an anti-PD-1 antibody, had a good activity against melanoma and other types of cancers. The toxicity profiles were tolerable. In the Keynote-028 phase Ib trial, pembrolizumab showed good clinical activity against recurrent or metastatic NPC. The overall response rate is 22%, and the disease control rate is 77.8%. This data is encouraging for further clinical trials of pembrolizumab for NPC.

PD-1/PD-L1 axis has an important role for the resistance of chemoradiation[18]. In patients refractory to chemoradiation, the expression of PD-1 and PD-L1 increased in the tumor. In animal model, sequential administration of anti-PD-1 after radiation significantly improved the progression free survival in mice with tumors [19]. This concept supports the investigator's sequential design for high-risk NPC patients.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent/assent for the trial.
2. Be more than 20 years of age on day of signing informed consent.
3. Have a performance status of 0 or 1 on the ECOG Performance Scale
4. Demonstrate adequate organ function as defined in Table 2

   * Hematological
   * Absolute neutrophil count (ANC) ≥1,500 /mcL
   * Platelets ≥100,000 / mcL
   * Hemoglobin ≥9 g/dL or ≥5.6 mmol/L without transfusion or EPO dependency (within 7 days of assessment)
   * Renal Serum creatinine OR Measured or calculateda creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≤1.5 X upper limit of normal (ULN) OR≥60 mL/min for subject with creatinine levels > 1.5 X institutional ULN
   * Hepatic
   * Serum total bilirubin ≤ 1.5 X ULN OR Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN
   * AST (SGOT) and ALT (SGPT)≤ 2.5 X ULN
   * Albumin >2.5 mg/dL
   * Coagulation
   * International Normalized Ratio (INR) or Prothrombin Time (PT)
   * Activated Partial Thromboplastin Time (aPTT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants ≤1.5 X ULN unless subject is receiving anticoagulant therapyas long as PT or PTT is within therapeutic range of intended use of anticoagulants aCreatinine clearance should be calculated per institutional standard.
5. Histology proven nasopharyngeal carcinoma. Biopsy at nasopharynx is mandatory.
6. Completing radiotherapy more than 66Gy (curative intent radiotherapy)
7. Detectable plasma EBV DNA: it is defined by the following criteria:

   1. The first test of plasma EBV DNA: 6-8 weeks after the last dose of radiotherapy.
   2. If the first test of plasma EBV DNA is detectable:

      * Within the "linear dynamic range": eligible by one single EBV DNA testing
      * Lower than the "linear dynamic range": it should be repeated within 2-4 weeks after the report day of first test of plasma EBV DNA. If both results are detectable, the patient is eligible
      * *The "linear dynamic range" is defined as the highest to the lowest quantifiable copy number established by means of a calibration curve (MIQE guidelines, 7.4.2 section, Clin Chem. 2009;55(4):611-22)
8. No detectable residual disease or distant metastases after imaging studies: The following examinations should be completed within 28 days after the report day of detectable plasma EBV DNA. If a repeated test of plasma EBV DNA is necessary by criteria 7, the following examination should be completed within 28 days after the report day of the repeated plasma EBV DNA test.

   1. For locally residual disease, head and neck MRI should be completed. For patients who cannot take MRI, CT scan with and without contrast should be completed.
   2. For distant metastases, one of the following studies should be completed.

      * Whole body PET-CT scan (if the modality is available)
      * CT scan with and without contrast of chest and abdomen, and bone scan
9. Female subject of childbearing potential should have a negative urine or serum pregnancy test. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
10. Female subjects of childbearing potential (Section 5.5.2) must be willing to use an adequate method of contraception as outlined in Section 5.5.2 - Contraception, for the course of the study through 120 days after the last dose of study medication. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
11. Male subjects of childbearing potential (Section 5.5.2) must agree to use an adequate method of contraception as outlined in Section 5.5.2- Contraception, starting with the first dose of study therapy through 120 days after the last dose of study therapy. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

Exclusion Criteria:

* The subject must be excluded from participating in the trial if the subject:

  1. Other malignancies diagnosed before or concurrently with the diagnosis of NPC.
  2. Take chemotherapy or other anti-cancer agents after curative chemoradiation.
  3. Documented residual / recurrent local disease or distant metastases after completing chemoradiation.
  4. Plasma EBV DNA is un-detectable.
  5. Unresolved grade 2 or more acute toxicities related to chemoradiation
  6. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
  7. Hypersensitivity to pembrolizumab or any of its excipients.
  8. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment. Topical or inhaled steroids is not considered as systemic treatment.
  9. Has known history of pneumonitis requiring steroids, or any evidence of active, non-infectious pneumonitis
  10. Has an active infection requiring systemic therapy 14 days before signing informed consent.
  11. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
  12. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
  13. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
  14. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
  15. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
  16. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
  17. Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-05-07 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
prolong one-year disease free survival (DFS-1y) | 5 years
  To examine the efficacy of pembrolizumab to prolong one-year disease free survival (DFS-1y) in nasopharyngeal carcinoma (NPC) patients with detectable plasma Epstein-Barr virus (EBV) DNA after curative chemoradiation.

CONTACTS AND LOCATIONS:
Overall Officials: Ruey-Long Hong, PhD, Principal Investigator — National Taiwan University Hospital
Locations (8):
- Taiwan (8):
  - Changhua Christian Hospital, Changhua
  - Chang Gung Memorial Hospital, Linkou District
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Koo Foundation Sun Yat-Sen Cancer Center, Taipei
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No